CLINICAL TRIAL: NCT04246255
Title: A New Method for Pain Relief, Intravenous Cannulation in Pediatric Patients; A Randomized Prospective Clinical Trial.
Brief Title: Pain Relief During Intravenous Cannulation in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Fatma Ferda Kartufan, Assistant Professor, MD, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KAEK 882
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cannula Site Pain; Local Anesthesia
Keywords: Local Anesthesia, Cannula Site Pain, Lidocaine Hydrocloride
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (Placebo Comparator): Serum Physiologic %0,9 ampules ; 0,3ml {spraying three times from a pump spray bottle that sprays 0,1 ml each time to Tegaderm + (2,5 cm x 4 cm) Non-Adherent Pad} 10 minutes before the IV cannula application
  Interventions: Drug: Placebo- Serum Fizyolojik Izotonik 0,9% 10 ml ampul
- Group L (Experimental): xylocaine %10 pump spray ; 30mg lidocaine {spraying three times from a pump spray bottle that sprays 0,1 ml each time to Tegaderm + (2,5 cm x 4 cm) Non-Adherent Pad} 10 minutes before the IV cannula application
  Interventions: Drug: Xylocaine 10% Oral

INTERVENTIONS:
Drug: Xylocaine 10% Oral — 50 ml of lidocaine solution maintained from xylocaine 10% oral that transferred to a bottle with a spray pump which pumps 0,1ml for each pump will be used for the experiment.
  3 pumps of lidocaine will be administrated to 3M TegadermTM +Pad Film Dressing with Non-Adherent Pad and put onto the skin for 10 minutes that IV cannula planned to be inserted.
  Other Names: EJACERA%10 sprey; LINCAINE sprey %10; LOCANEST sprey %10; PRECOXIN %10 sprey; VEMCAINE pump sprey %10
  Arms: Group L
Drug: Placebo- Serum Fizyolojik Izotonik 0,9% 10 ml ampul — 50 ml of Serum physiologic in a bottle with a spray pump which pumps 0,1ml for each pump will be used for placebo.
  3 pumps of placebo will be administrated to 3M TegadermTM +Pad Film Dressing with Non-Adherent Pad and put onto the skin for 10 minutes that IV cannula planned to be inserted.
  Other Names: Serum Fizyolojik Onfarma 10 Ml, 10 Ampul,; Serum Fizyolojik İzotonik %0,9 10 Ml, 100 Ampul; Serum Fizyolojik Biofarma % 0,9, 10 Ml 100 Ampul
  Arms: Group C

SUMMARY:
Performing intravenous (IV) cannulation to pediatric patients might be much harder than adult ones according to their anxiety levels. However, managing adult patients during intravenous cannulation is also challenging if he or she had a noxious memory about the situation or has a low pain threshold. Therefore, it is essential to relieve the pain of an IV needle or an IV cannula insertion in the pediatric patient population. Lidocaine Hcl spray (Xylocaine 10% Oral ) will be utilized to the research group, and Serum Physiologic (Serum Fizyolojik %0,9 10 ml ampule, Biofarma İlaç San. ve Tic A.Ş., İstanbul, Turkey) will be utilized to the control group of the study. Both medications will be administrated by spraying the formula three times to an adhesive bandage and placing it to the skin that IV cannulation will be performed. After waiting for a minimum of 5 to a maximum of 15 minutes ( waiting time is closely associated with the patient's anxiety level), IV cannulation will be performed from the same area by an experienced pediatric nurse. The investigator hypothesizes that utilizing the spray form of the Lidocaine Hcl formula to the skin with an adhesive bandage before IV cannulation might lower the pain of the manipulation in pediatric patients, which might cause lower anxiety levels with stable vital signs.

DETAILED DESCRIPTION:
The G-Power 3.0.10. Computed required sample size (alpha:0.05, effect size:0.3 and power 0.8) related to t-test of the difference between two dependent means(matched pairs) according to the 5% change of before and after heartbeat outcome parameters with Standard derivations of ( -/+12 to +/-15). The total sample size of ninety participants is evaluated to be enough for the study. However, fifty participants are planned to be enrolled in each group (a total of 100 participants) to compensate for possible losses in this prospective, randomized clinical study. Six parameters will be evaluated, and three scales will be performed in each group. The six parameters are Heart Rate-1, Spo2-1, Body Temperature-1, Heart Rate-2, Spo2-2, Body Temperature-2. The three scales are 11 point Verbal Numeric Rating Scale-1, 11 point Verbal Numeric Rating Scale-2, and Visual Analog Scale. Those parameters will be measured non-invasively, without causing any pain.

The randomization is planned to be done with the sealed envelope modeling. One of the envelopes is planned to be chosen by each participant after the written consent form approval from the child and his/her parents. The envelopes have either a "C" letter or "L" letter inside representing C as {Group C: "The Control Group"}, representing L as {Group L: "The Lidocaine Group"} will be opened by the principal investigator. The bottle 1(Serum Physiologic inside) or bottle 2( Lidocaine inside) will be given to the ward nurse according to the letters in the envelope. The ward nurse will be blinded according to the ingredients in the bottles. The outcome parameters and the scales will be recorded by the nurse in the investigation. The nurse in the investigation will be blinded about the groups, the envelopes and the ingredients performed to the participants.

The study is planned to last in 4 months (16 weeks) time. However, in the middle of the study( 25 participants undertaken within each group), post-doc tests are planned to be done. If the power of the study according to the post-Hoc tests are more than 80%, the study will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* The subject has to be treated with any drug submitted via intravenous cannula.
* The subject weighted more than 10 kg.
* The subject has a maximum ASA-2 score.

Exclusion Criteria:

* Allergic to amide group local anesthetics.
* The subject has a dermatological disease.

Ages: 72 Months to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Heart Rate-1 | It is going to be measured in the first minute(1st min) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Heart Beat per minute, data obtained from SpO2 pediatric probe, before IV cannula insertion
SpO2-1 | It is going to be measured in the first minute(1st min) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Peripheral Oxygen concentration, data obtained from SpO2 pediatric probe, before IV cannula insertion.
Body Temperature-1 | It is going to be measured in the second minute(2nd min) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Body temperature, data obtained from tympanic temperature, before IV cannula insertion
Heart Rate-2 | It is going to be measured in the last 5 minutes period of the study(approximately in the 12th minute) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Heart Beat per minute, data obtained from SpO2 pediatric probe, after IV cannula insertion
SpO2-2 | It is going to be measured in the last 5 minutes period of the study(approximately in the 12th minute) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Peripheral Oxygen concentration, data obtained from SpO2 pediatric probe, after IV cannula insertion.
Body Temperature-2 | It is going to be measured in the last 5 minutes period of the study(approximately in the 13th minute) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  Body temperature, data obtained from tympanic temperature, after IV cannula insertion

SECONDARY OUTCOMES:
11-point Verbal Numeric Rating Scale-1 (VNS-1) | It is going to be measured in the third minute(3rd min) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  The subject is going to be asked to rate the cannula insertion pain, which the subject had experienced before the study ( if they had no experience Outcome 7 would stay empty), verbally according to the intensity from 0-10 with 0 representing "no pain" and 10 representing "the most intense pain imaginable."
Visual Analog Scales | It is going to be measured in the in the last 5 minutes period of the study(approximately in the 14th minute) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  The subject will be asked to rate the cannula insertion pain after insertion by placing a vertical mark on a 100 mm horizontal VAS. The left and right extremes of the VAS are labeled as; "least possible pain" and "worst possible pain" respectively. 100mm VAS is devided into 5 categorical descriptors: "much less pain," "a little less pain," "about the same pain," "a little more pain," or "much more pain."
11-point Verbal Numeric Rating Scale-2 (VNS-2) | It is going to be measured in the in the last 5 minutes period of the study(approximately in the 15th minute) of the total 15 mins. study, for each participant, through study completion up to 16 weeks.
  The subject is going to be asked to rate the cannula insertion pain after insertion verbally according to the intensity from 0-10 with 0 representing "no pain" and 10 representing "the most intense pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Ferda F Kartufan, Asst.Prof., Principal Investigator — Yeditepe University Anesthesiology and Reanimation Department
Locations (1):
- Yeditepe University, Istanbul, İçerenköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cozzi G, Borrometi F, Benini F, Neri E, Rusalen F, Celentano L, Zanon D, Schreiber S, Ronfani L, Barbi E. First-time success with needle procedures was higher with a warm lidocaine and tetracaine patch than an eutectic mixture of lidocaine and prilocaine cream. Acta Paediatr. 2017 May;106(5):773-778. doi: 10.1111/apa.13764. Epub 2017 Feb 21. PMID 28130888
- [Background] Kim WO, Song BM, Kil HK. Efficacy and safety of a lidocaine/tetracaine medicated patch or peel for dermatologic procedures: a meta-analysis. Korean J Anesthesiol. 2012 May;62(5):435-40. doi: 10.4097/kjae.2012.62.5.435. Epub 2012 May 24. PMID 22679540